CLINICAL TRIAL: NCT01219452
Title: Effects of Intramuscular Injection of Umbilical Cord Mesenchymal Stem Cell on the Ventricular Function of Children With Idiopathic Dilated Cardiomyopathy
Brief Title: Intramuscular Injection of Mesenchymal Stem Cell for Treatment of Children With Idiopathic Dilated Cardiomyopathy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qingdao University (Other)
Responsible Party: Qingdao University, Organization: Stem Cell Research Center of Medical School Hospital of Qingdao University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSCKX002
Record Dates: First submitted 2010-10-12; First posted 2010-10-13 (Estimated); Last update posted 2010-10-28 (Estimated); Status verified 2010-05

CONDITIONS: Dilated Cardiomyopathy
Keywords: Dilated Cardiomyopathy; Umbilical cord; Mesenchymal stem cells; Children
MeSH Terms: conditions — Cardiomyopathy, Dilated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- umbilical cord mesenchymal stem cells (Experimental): intramuscular injection of umbilical cord mesenchymal stem cell
  Interventions: Biological: umbilical cord mesenchymal stem cells

INTERVENTIONS:
Biological: umbilical cord mesenchymal stem cells — Multiple intra muscular injection of mesenchymal stem cells derived from human umbilical cord.
  Other Names: mesenchymal stem cells

SUMMARY:
The main aim of the study is to determine whether intramuscular injection of umbilical cord mesenchymal stem cells can improve the ventricular function of children with idiopathic dilated cardiomyopathy(IDCM); Secondary end-points will be: 1)To explore the possible mechanism of the improvement of ventricular function in children with IDCM and 2) to evaluate the safety of intramuscular injection of umbilical cord mesenchymal stem cell.

DETAILED DESCRIPTION:
Children with Idiopathic dilated cardiomyopathy class II to III NYHA with ejection fraction over 20% were selected for phase II clinical trial, umbilical cord mesenchymal stem cells were injected into limb muscle and followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Children of both genders with established clinical and echocardiographic diagnosis of dilated cardiomyopathy whose parents accept to participate in the trail.
* They should have symptoms and /or signs of heart failure, despite optimized medical treatment.
* Ejection fraction of left ventricular should be less than 50%, but more than 20%.

Exclusion Criteria:

* associate coronary artery disease.
* any history or suspicion of a toxic , pharmacologic or deposit etiology.
* associated malignant or pre -malignant systemic disease.
* associated hematologic disorder.
* a history of sustained ventricular tachycardia or fibrillation.
* a history of syncope during the previous year, or with an active infectious disease or positive tests to viral disease.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-11 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
echocardiography | 3 months

SECONDARY OUTCOMES:
24h HOLTER | 2 months
The level of serum BNP,TNI,HGF、LIF and G/M-CSF | 3 months
The expression level of c-kit,CD31,CD133 on peripheral blood mononuclear cells | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: zipu li, MD Phd, Study Director — The Affiliated Hospital of Qingdao University
Locations (1):
- Stem Cell Research Center of Medical School Hospital of Qingdao University, Qingdao, Shandong, China